CLINICAL TRIAL: NCT06430814
Title: Clinical Biomarker of Paclitaxel-induced Peripheral Neuropathy
Status: Recruiting | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Sygehus Lillebaelt (Other); Sonderborg Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AKF-403
Record Dates: First submitted 2024-04-25; First posted 2024-05-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators are taking blood samples to analyze the NFL level, paclitaxel concentration, and looking at DNA sequencing associated with PIPN. The investigators will also take skin biopsies to look at the nerve fiber density and if gene and protein expression of relevant genes changes following paclitaxel treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breastcancer patients: A total of 188 patients diagnosed with breast cancer who are scheduled for paclitaxel treatment, either as adjuvant or neo-adjuvant treatment, will be recruited across three trial sites.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Investigation of which patients treated with paclitaxel have an increased risk of developing peripheral neuropathy.

DETAILED DESCRIPTION:
The primary aim of this study is to validate the protein neurofilament light chain (NFL) as a biomarker of the side effect paclitaxel-induced peripheral neuropathy (PIPN) and its utility in predicting this side effect in patients with breast cancer. The investigators want to include 188 patients at four different trial sites. The patients must follow their normal treatment cycles while getting blood drawn during their treatment period however maximal 4 cycles.

Blood samples are dawn before treatment initiation and once before each new cycle start in order to measure neurofilament light chain (NFL) before and during treatment. The investigators also want to take a skin biopsy before treatment start and after either cycle 3 or 4.

The primary endpoint of the study is if serum NFL>100 pg/ml after first cycle of paclitaxel can predict early termination of paclitaxel due to peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Willing to give informed consent
* Scheduled to receive neo-adjuvant or adjuvant paclitaxel treatment
* Able to speak and understand Danish
* Diagnosed with breast cancer
* Paclitaxel naïve patients

Exclusion Criteria:

* Neurodegenerative diseases (e.g., neuropathy from another cause, previous apoplexy, disc herniation
* Type 1 or 2 diabetes
* Pregnant
* Breastfeeding
* Relapse of cancer diagnosis
* Diagnosed with human immunodeficiency virus (HIV)
* Participation in other clinical trials where the dose of paclitaxel is changed, or the aim is to prevent neuropathic pain or decrease NFL level (except if the intervention is to use cooling gloves).
* Previous treatment with neurotoxic chemotherapy
* Chronic pain from another cause
* Metastatic cancer

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: A total of 188 patients diagnosed with breast cancer who are scheduled for paclitaxel treatment, either as adjuvant or neo-adjuvant treatment, will be recruited across four trial sites.
Sampling Method: Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
NFL level correlation | Before treatment start and during four cycles (one cycle equals 3 weeks)
  The primary endpoint of the study is if serum NFL>100 pg/ml after first cycle (one cycle equals 3 weeks) of paclitaxel can predict early termination of paclitaxel due to peripheral neuropathy.

SECONDARY OUTCOMES:
Paclitaxel exposure | Before treatment start and during four cycles (one cycle equals 3 weeks)
  To measure if high concentration of paclitaxel exposure is correlated to high NFL level in blood
Genes and PIPN | Before treatment start and during four cycles (one cycle equals 3 weeks)
  To measure if genetic variants in genes (e.g., CYP2C8*3, EPHA4/5, FGD4) are associated with more server PIPN symptoms.
Genes and NFL | Before treatment start and during four cycles (one cycle equals 3 weeks)
  To measure if genetic variants in genes (e.g., CYP2C8*3, EPHA4/5, FGD4) are associated with high NFL concentration in blood.
Genes and Paclitaxel | Before treatment start and during four cycles (one cycle equals 3 weeks)
  To measure if genetic variants in genes (e.g., CYP2C8*3, EPHA4/5, FGD4) are associated with high paclitaxel concentration in blood.
Drug-drug interactions | Before treatment start and during four cycles (one cycle equals 3 weeks)
  Investigate if and which specific drug-drug interactions are correlated to developing PIPN.
Skin biopsies | Before treatment start and during four cycles (one cycle equals 3 weeks)
  Obtain skin biopsies from patients to elucidate which molecular mechanisms and phenotypes are associated with PIPN.
IENFD | Before treatment start and during four cycles (one cycle equals 3 weeks)
  Obtain skin biopsies at baseline and at the beginning of cycle 3 or 4 (one cycle equals 3 weeks) to assess if the intraepidermal nerve fiber density (IENFD) changes during paclitaxel treatment.
PHS | Before treatment start and during four cycles (one cycle equals 3 weeks)
  To assess whether the patients who have a sensation of heat during cooling of the skin (PHS) are also those who experience neuropathic pain.
Nerve fiber dysfunction | Before treatment start and during four cycles (one cycle equals 3 weeks)
  To examine if increased NFL level is correlated to changes in small and large nerve fibers dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Bork Iversen, Study Chair — University of Southern Denmark
Locations (3):
- Denmark (3):
  - Odense University Hospital, Odense
  - University Hospital of Southern Denmark, Sønderborg, Sønderborg
  - University Hospital of Southern Denmark, Vejle, Vejle

IPD SHARING:
Plan to Share IPD: No
Data on individual participants is not allowed due to GDPR